CLINICAL TRIAL: NCT04659863
Title: Two Part (Double-blind Inclisiran Versus Placebo [Year 1] Followed by Open-label Inclisiran [Year 2]) Randomized Multicenter Study to Evaluate Safety, Tolerability, and Efficacy of Inclisiran in Adolescents (12 to Less Than 18 Years) With Homozygous Familial Hypercholesterolemia and Elevated LDL-cholesterol (ORION-13)
Brief Title: Study to Evaluate Efficacy and Safety of Inclisiran in Adolescents With Homozygous Familial Hypercholesterolemia
Acronym: ORION-13
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKJX839C12302; 2020-002755-38 (EudraCT Number)
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Familial Hypercholesterolemia - Homozygous
Keywords: Homozygous familial hypercholesterolemia (HoFH); LDL-cholesterol (LDL-C); adolescents; pediatric; small interfering ribonucleic acid (siRNA)
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — ALN-PCS; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel (Year 1) to single-group (Year 2)
Who Masked: Participant, Investigator
Masking Description: Masked (Year 1) to No Masking (Year 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 - Inclisiran (Experimental): Inclisiran sodium 300 mg subcutaneous (sc) injection (given at Days 1, 90 and 270)
  Interventions: Drug: Inclisiran
- Part 1 - Placebo (Placebo Comparator): Placebo sc injection (given at Day 1, 90 and 270)
  Interventions: Drug: Placebo
- Part 2 - Inclisiran (Total) (Experimental): Inclisiran sodium 300 mg sc injection (given at Days 450 and 630). In addition, participants assigned to placebo in Part 1 received inclisiran sodium 300 mg sc injection on Day 360, while participants assigned to inclisiran in Part 1 received placebo sc injection on Day 360.
  Interventions: Drug: Inclisiran

INTERVENTIONS:
Drug: Inclisiran — Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) in 1.5 mL solution for subcutaneous injection
  Other Names: KJX839
  Arms: Part 1 - Inclisiran; Part 2 - Inclisiran (Total)
Drug: Placebo — Sterile normal saline (0.9% sodium chloride in water for injection) for subcutaneous injection
  Other Names: Saline solution
  Arms: Part 1 - Placebo

SUMMARY:
This was a pivotal phase III study designed to evaluate safety, tolerability, and efficacy of inclisiran in adolescents with homozygous familial hypercholesterolemia (HoFH) and elevated low density lipoprotein cholesterol (LDL-C).

DETAILED DESCRIPTION:
This was a two-part (double-blind, inclisiran versus placebo [Year 1] followed by open-label inclisiran [Year 2]) multicenter study in adolescents (aged 12 to < 18 years) with HoFH and elevated LDL-C (> 130 mg/dL; 3.4 mmol/L) on stable, individualized, optimal standard of care (SoC) background lipid-lowering therapy (including maximally tolerated statin treatment, at the Investigator's discretion) to evaluate the safety, tolerability, and efficacy of inclisiran in this pediatric patient population.

Following an approximately 4-week screening/run-in period, the study had 2 sequential parts as follows:

Part 1/Year 1: 12 months double-blind, parallel group period, in which participants were randomized in a 2:1 ratio to receive either inclisiran sodium 300 mg subcutaneous (s.c.) or placebo. The primary endpoint was assessed at Day 330.

Part 2/Year 2: 12 months single arm, open-label follow-up period, with all participants receiving inclisiran sodium 300 mg s.c.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous Familial Hypercholesterolemia (HoFH) diagnosed by genetic confirmation
* Fasting LDL-C >130 mg/dL (3.4 mmol/L) at screening
* On maximally tolerated dose of statin (investigator's discretion) with or without other lipid-lowering therapy; stable for ≥ 30 days before screening
* Male or female participants >=12 to <18 years of age at screening

Exclusion Criteria:

* Documented evidence of a null (negative) mutation in both LDLR alleles
* Heterozygous familial hypercholesterolemia (HeFH)
* Active liver disease
* Secondary hypercholesterolemia, e.g. hypothyroidism or nephrotic syndrome
* Previous treatment with monoclonal antibodies directed towards PCSK9 (within 90 days of screening)
* Treatment with mipomersen or lomitapide (within 5 months of screening)
* Recent and/or planned use of other investigational medicinal products or devices

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Excel Medical Clinical Trials LLC, Boca Raton, Florida, United States
- Novartis Investigative Site, Québec, Quebec, Canada
- Novartis Investigative Site, Bron, France
- Greece (2):
  - University General Hospital of Ioannina, Ioannina, GR
  - Metropolitan Hospital, Athens
- Lebanon (2):
  - American University of Beirut Medical Center, Beirut
  - Hotel Dieu de France Hospital, El Achrafiyé
- Novartis Investigative Site, Kuala Lumpur, Malaysia
- Novartis Investigative Site, Amsterdam, Netherlands
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wiegman A, Peterson AL, Hegele RA, Bruckert E, Schweizer A, Lesogor A, Wang Y, Defesche J. Efficacy and Safety of Inclisiran in Adolescents With Genetically Confirmed Homozygous Familial Hypercholesterolemia: Results From the Double-Blind, Placebo-Controlled Part of the ORION-13 Randomized Trial. Circulation. 2025 Jun 24;151(25):1758-1766. doi: 10.1161/CIRCULATIONAHA.124.073233. Epub 2025 May 20. PMID 40391436
- [Derived] Reijman MD, Schweizer A, Peterson ALH, Bruckert E, Stratz C, Defesche JC, Hegele RA, Wiegman A. Rationale and design of two trials assessing the efficacy, safety, and tolerability of inclisiran in adolescents with homozygous and heterozygous familial hypercholesterolaemia. Eur J Prev Cardiol. 2022 Jul 20;29(9):1361-1368. doi: 10.1093/eurjpc/zwac025. PMID 35175352
- [Derived] Warden BA, Duell PB. Inclisiran: A Novel Agent for Lowering Apolipoprotein B-containing Lipoproteins. J Cardiovasc Pharmacol. 2021 Aug 1;78(2):e157-e174. doi: 10.1097/FJC.0000000000001053. PMID 33990512
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2616
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=696

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen participants were randomized from 9 study centers in 8 countries. The breakdown of countries and study centers for the randomized participants was as follows: Canada (1), France (1), Greece (1), Lebanon (1), Malaysia (1), Netherlands (1), Turkey (2), and United States (1).
Pre-assignment Details: The study had an approximately 4-week screening/run-in period
Groups:
- Part 1- Inclisiran: Inclisiran sodium 300 mg subcutaneous (sc) injection (given at Days 1, 90 and 270)
Period: Part 1 (Double-blind Period)
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Started | 9 | 4 | 0
Completed | 9 | 4 | 0
Not Completed | 0 | 0 | 0
Period: Part 2 (Open-label Period)
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Started | 0 | 0 | 13
Completed | 0 | 0 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics are based on all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 4 | 13
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.54) | 15.1 (2.66) | 14.8 (1.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  White | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in LDL-C From Baseline to Day 330 (Part 1/Year 1)
Description: Percentage change in low-density lipoprotein cholesterol (LDL-C) from baseline to Day 330 (Year 1)
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization.
Measure: Mean (Standard Deviation); unit: percent change in LDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 9 | 4
percent change in LDL-C | -21.6 (13.36) | 11.7 (30.52)
Statistical Analysis 1: Comparison: Part 1- Inclisiran vs Part 1 - Placebo; Test type: Other; Mean Difference (Net) = -33.25, 95% CI 2-sided [-59.17 to -7.34]

2. Secondary Outcome: Time-adjusted Percent Change in LDL-C From Baseline After Day 90 and up to Day 330 (Part 1/Year 1)
Description: Time-adjusted percent change in LDL-C (after Day 90 and up to Day 330), calculated as the average of percent changes from baseline to Days 150, 270 and 330
Time Frame: Baseline, after Day 90 up to Day 330
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Time-adjusted percent change in LDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 9 | 4
Time-adjusted percent change in LDL-C | -21.0 (15.11) | 13.0 (41.88)

3. Secondary Outcome: Percent Change in LDL-C From Baseline up to Day 720
Description: Percentage change in LDL-C from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Percent change in LDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
Percent change in LDL-C
  Day 90: number analyzed (Participants) | 9 | 4 | 0
  Day 90 | -26.1 (13.53) | 6.8 (16.83) |
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -24.1 (14.65) | 17.0 (41.22) |
  Day 270: number analyzed (Participants) | 9 | 4 | 0
  Day 270 | -17.3 (21.64) | 10.2 (54.00) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -21.6 (13.36) | 11.7 (30.52) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -19.3 (14.75) | 5.4 (28.24) |
  Day 450: number analyzed (Participants) | 0 | 0 | 13
  Day 450 |  |  | -11.0 (25.28)
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -12.5 (22.52)
  Day 630: number analyzed (Participants) | 0 | 0 | 13
  Day 630 |  |  | -9.4 (26.16)
  Day 720: number analyzed (Participants) | 0 | 0 | 13
  Day 720 |  |  | -12.6 (28.45)

4. Secondary Outcome: Absolute Change in LDL-C From Baseline up to Day 720
Description: Absolute change in LDL-C from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
mg/dL
  Day 90: number analyzed (Participants) | 9 | 4 | 0
  Day 90 | -70.6 (48.81) | 16.5 (44.96) |
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -66.1 (61.85) | 20.3 (91.34) |
  Day 270: number analyzed (Participants) | 9 | 4 | 0
  Day 270 | -47.1 (83.15) | -9.3 (134.14) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -62.9 (52.35) | 11.8 (69.94) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -50.8 (44.65) | -4.3 (69.84) |
  Day 450: number analyzed (Participants) | 0 | 0 | 13
  Day 450 |  |  | -36.6 (75.08)
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -46.8 (73.04)
  Day 630: number analyzed (Participants) | 0 | 0 | 13
  Day 630 |  |  | -41.9 (92.47)
  Day 720: number analyzed (Participants) | 0 | 0 | 13
  Day 720 |  |  | -39.8 (96.59)

5. Secondary Outcome: Percent Change in Apo B From Baseline up to Day 720
Description: Percentage change in apolipoprotein B (Apo B) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Percent change in Apo B
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
Percent change in Apo B
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -20.3 (12.92) | 10.0 (27.05) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -18.5 (10.47) | 4.5 (17.91) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -14.8 (10.11) | 10.6 (21.33) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -5.7 (25.96)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -7.3 (29.36)

6. Secondary Outcome: Absolute Change in Apo B From Baseline up to Day 720
Description: Absolute change in apolipoprotein B (Apo B) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
mg/dL
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -37.3 (33.35) | 7.5 (48.72) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -35.8 (30.33) | 0.3 (35.85) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -28.7 (27.16) | 12.0 (32.89) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -18.8 (45.81)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -19.6 (51.64)

7. Secondary Outcome: Percent Change in Lp(a) From Baseline up to Day 720
Description: Percentage change in lipoprotein (a) [Lp(a)] from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Percent change in Lp(a)
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
Percent change in Lp(a)
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -0.7 (24.81) | -4.4 (9.20) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -0.3 (21.27) | -16.5 (27.29) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -1.7 (16.57) | -12.1 (31.51) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -7.2 (31.39)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -8.8 (22.03)

8. Secondary Outcome: Absolute Change in Lp(a) From Baseline up to Day 720
Description: Absolute change in lipoprotein (a) [Lp(a)] from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
nmol/L
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | 8.9 (28.41) | -0.3 (1.26) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | 2.8 (15.01) | 5.3 (15.86) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | 5.8 (7.03) | 0.5 (9.75) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | 3.0 (14.45)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -0.3 (9.12)

9. Secondary Outcome: Percent Change in Non-HDL-C From Baseline up to Day 720
Description: Percentage change in non-high density lipoprotein cholesterol (non-HDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Percent change in non-HDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
Percent change in non-HDL-C
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -24.0 (13.83) | 19.0 (43.34) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -23.3 (10.99) | 9.4 (34.93) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -20.1 (10.91) | 7.1 (24.38) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -11.8 (25.33)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -13.0 (23.65)

10. Secondary Outcome: Absolute Change in Non-HDL-C From Baseline up to Day 720
Description: Absolute change in non-high density lipoprotein cholesterol (non-HDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
mg/dL
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -73.8 (68.01) | 28.8 (94.01) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -74.4 (57.63) | 4.3 (82.16) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -60.0 (44.74) | 6.0 (56.11) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -51.4 (81.53)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -45.8 (89.10)

11. Secondary Outcome: Percent Change in Total Cholesterol From Baseline up to Day 720
Description: Percentage change in total cholesterol from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Percent change in total cholesterol
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
Percent change in total cholesterol
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -19.0 (12.49) | 16.0 (37.96) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -19.1 (10.30) | 8.7 (30.54) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -16.1 (9.53) | 6.8 (21.06) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -9.3 (20.73)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -9.6 (20.86)

12. Secondary Outcome: Absolute Change in Total Cholesterol From Baseline up to Day 720
Description: Absolute change in total cholesterol from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
mg/dL
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -69.7 (67.42) | 29.5 (99.30) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -71.4 (56.65) | 8.8 (84.68) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -57.3 (43.82) | 10.0 (59.14) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -46.5 (80.87)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -40.4 (88.44)

13. Secondary Outcome: Percent Change in Triglycerides From Baseline up to Day 720
Description: Percentage change in triglycerides from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Percent change in triglycerides
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
Percent change in triglycerides
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | 0.3 (31.92) | -15.7 (5.97) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -9.6 (30.66) | -5.8 (31.90) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | 11.4 (24.72) | 14.1 (54.93) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | 4.7 (37.21)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | 2.9 (26.02)

14. Secondary Outcome: Absolute Change in Triglycerides From Baseline up to Day 720
Description: Absolute change in triglycerides from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
mg/dL
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -3.4 (23.80) | -15.0 (7.53) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -9.4 (21.98) | -2.3 (25.01) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | 8.7 (24.15) | 28.0 (72.23) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | 3.3 (34.32)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | 3.9 (27.40)

15. Secondary Outcome: Percent Change in HDL-C From Baseline up to Day 720
Description: Percentage change in high density lipoprotein cholesterol (HDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Percent change in HDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
Percent change in HDL-C
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | 10.0 (13.22) | -0.1 (20.06) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | 7.5 (12.93) | 10.9 (12.48) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | 6.7 (20.60) | 9.2 (21.20) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | 12.3 (17.63)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | 13.9 (18.81)

16. Secondary Outcome: Absolute Change in HDL-C From Baseline up to Day 720
Description: Absolute change in high density lipoprotein cholesterol (HDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
mg/dL
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | 4.1 (5.18) | 0.8 (7.50) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | 3.0 (5.05) | 4.5 (5.07) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | 2.7 (7.75) | 4.0 (8.76) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | 4.9 (7.94)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | 5.4 (7.81)

17. Secondary Outcome: Percent Change in VLDL-C From Baseline up to Day 720
Description: Percentage change in very low density lipoprotein cholesterol (VLDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Percent change in VLDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
Percent change in VLDL-C
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -7.0 (70.31) | 74.5 (108.97) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -29.0 (49.96) | 2.0 (113.44) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -17.0 (60.36) | 34.6 (56.37) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | 9.5 (98.44)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -1.4 (69.03)

18. Secondary Outcome: Absolut Change in VLDL-C From Baseline up to Day 720
Description: Absolute change in very low density lipoprotein cholesterol (VLDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
mg/dL
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -7.7 (11.39) | 8.5 (20.37) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -11.6 (11.71) | -7.5 (18.21) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -9.2 (17.89) | 10.3 (21.00) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -4.6 (18.41)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -6.0 (18.81)

19. Secondary Outcome: Percent Change in Apo A1 From Baseline up to Day 720
Description: Percentage change in apolipoprotein A1 (Apo A1) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Percent change in Apo A1
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
Percent change in Apo A1
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -0.9 (10.72) | -1.3 (2.27) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -2.1 (10.87) | 9.0 (7.02) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | 3.1 (16.49) | 13.7 (12.99) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | 12.8 (12.08)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | 6.5 (10.10)

20. Secondary Outcome: Absolute Change in Apo A1 From Baseline up to Day 720
Description: Absolute change in apolipoprotein A1 (Apo A1) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
mg/dL
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -1.2 (14.10) | -1.3 (2.36) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -2.7 (13.47) | 10.3 (7.41) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | 4.2 (18.82) | 16.0 (14.79) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | 14.9 (13.25)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | 7.4 (12.40)

21. Secondary Outcome: Percent Change in PCSK9 From Baseline up to Day 720
Description: Percentage change in proprotein convertase subtilisin/kexin type 9 (PCSK9) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: Percent change in PCSK9
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
Percent change in PCSK9
  Day 90: number analyzed (Participants) | 9 | 4 | 0
  Day 90 | -56.8 (13.73) | -17.3 (14.77) |
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -60.4 (12.62) | -1.7 (11.11) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -65.3 (12.51) | -5.1 (19.60) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -59.7 (9.05) | -2.8 (22.65) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -68.1 (10.57)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -64.1 (12.12)

22. Secondary Outcome: Absolut Change in PCSK9 From Baseline up to Day 720
Description: Absolute change in proprotein convertase subtilisin/kexin type 9 (PCSK9) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 9 | 4 | 13
ng/mL
  Day 90: number analyzed (Participants) | 9 | 4 | 0
  Day 90 | -278.7 (113.31) | -98.5 (87.46) |
  Day 150: number analyzed (Participants) | 9 | 4 | 0
  Day 150 | -296.3 (118.18) | -6.1 (64.82) |
  Day 330: number analyzed (Participants) | 9 | 4 | 0
  Day 330 | -323.1 (129.32) | -35.3 (100.97) |
  Day 360: number analyzed (Participants) | 9 | 4 | 0
  Day 360 | -292.6 (100.44) | -14.0 (127.42) |
  Day 510: number analyzed (Participants) | 0 | 0 | 13
  Day 510 |  |  | -347.3 (106.3)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 13
  Day 720 (study completion) |  |  | -327.7 (110.4)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 90 days post treatment or 30 days after last study visit, whichever was longer, up to a maximum duration of approximately 2 years.
Groups:
- Part 1 - Inclisiran: Inclisiran sodium 300 mg subcutaneous injection (given at Days 1, 90 and 270)
- Part 1 - Placebo: Placebo subcutaneous injection (given at Day 1, 90 and 270)
- Part 2 - Inclisiran (Total): Inclisiran sodium 300 mg subcutaneous injection (given at Days 450 and 630). In addition, participants assigned to placebo in Part 1 received inclisiran sodium 300 mg sc injection on Day 360, while participants assigned to inclisiran in Part 1 received placebo sc injection on Day 360
Arm/Group | Part 1 - Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/4 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/4 | 0/13
Other Adverse Events (participants affected / at risk) | 7/9 | 1/4 | 8/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Inclisiran (N=9) | Part 1 - Placebo (N=4) | Part 2 - Inclisiran (Total) (N=13)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 1
Injection site erythema (General disorders) | 1 | 0 | 1
Injection site reaction (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
COVID-19 (Infections and infestations) | 4 | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Carotid intima-media thickness increased (Investigations) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Xanthoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT04659863/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT04659863/SAP_001.pdf